CLINICAL TRIAL: NCT01226134
Title: Effect Of Itopride On Gastric Emptying And Accommodation In Patients With Functional Dyspepsia
Acronym: EIGEAPFD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Dr. Shahab Abid, Aga Khan University,Karachi, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 965-Med/ERC-08
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-07

CONDITIONS: Functional Dyspepsia; Gastric Emptying; Gastric Accommodation
Keywords: Functional Dyspepsia; Itopride; Gastric Emptying; Gastric Accommodation; Dyspeptic Symptoms
MeSH Terms: interventions — itopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.Itopride Group (Experimental): The itopride group will receive itopride 150mg per day(50mg TDS)for four weeks
  Interventions: Drug: Itopride,
- 2.Control placebo group (Placebo Comparator): The control group will receive placebo tablets for four weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itopride, — Itopride,50 mg capsules,thrice a day,for Four weeks
  Other Names: Gananton
  Arms: 1.Itopride Group
Drug: Placebo — placebo capsules,thrice a day for four weeks
  Arms: 2.Control placebo group

SUMMARY:
Pathogenesis of functional dyspepsia is poorly understood. Gastrointestinal motor abnormalities, Helicobacter pylori infection, impaired gastric accommodation to a meal, hypersensitivity of the afferent nerves of the gut, psychological disturbances and central nervous system dysfunction have been proposed.

Pharmacological treatments for patients with functional dyspepsia remain unsatisfactory. Only small benefits relative to placebo have been found with histamine H2 receptor antagonists, proton pump inhibitor and Helicobacter pylori eradication.

Itopride is a dopamine antagonist with acetylcholinesterase inhibitory actions. This agent is currently indicated for patients with various upper GI symptoms.

This study is aimed to evaluate the effect of Itopride on gastric emptying(by 13-C Octanoic acid breath Test), accommodation (by Gastric Scintigraphy SPECT and slow nutrient drinking test)and symptoms in FD patients

DETAILED DESCRIPTION:
phase3 clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. All adult male or non-pregnant female patients who are diagnosed as functional dyspepsia and fulfilling Rome III criteria (1) will be considered
2. Patients should be negative for H. pylori on gastric biopsy and Urea Breath Test.
3. duodenal biopsy in these patients should be negative for giardiasis or celiac disease or any other established organic pathology
4. A normal upper abdominal ultrasound
5. Willing to participate and give consent for participation in the study.

Exclusion Criteria:

1. Age <18 years
2. Helicobacter Pylori positive on gastric biopsy and / or UBT.
3. Taking other medications that alter gastric motility like macrolide

   * anti-emetics and antibiotics .
4. Pregnant or breast-feeding females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-03 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of Itopride on Gastric Emptying,accommodation and capacity of tolerating a nutrient drink in patients with Functional Dyspepsia | 18 months

SECONDARY OUTCOMES:
To assess the effect of Itopride on symptom improvement in patient with Functional Dyspepsia | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Abid, MD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan